CLINICAL TRIAL: NCT05983848
Title: An Observational Study Exploring the Value 99mMaracticaltide Imaging for Predicting Outcomes for Patients With Rheumatoid Arthritis Undergoing Tapering of Therapy
Brief Title: Scintigraphy for Prediction In Rheumatoid Intentional Therapy Tapering
Acronym: SPIRITT
Status: Not yet recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other); Serac Healthcare (Unknown); Versus Arthritis (Other)
Responsible Party: Sponsor
Other Study IDs: 825832
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Additional study bloods (20ml) will be taken at baseline and 6-month visits for serological markers of inflammation and neoangiogenesis. Serum samples will be given a trial ID and stored in the Infectious Disease Biobank, King's College London. Samples will be processed, stored and disposed in accordance with all applicable legal and regulatory requirements, including the Human Tissue Act 2004 and any amendments thereafter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: 99mMaracticaltide imaging — 7.3.1 99mTc-maraciclatide imaging This will be undertaken at baseline and optionally at 8-12 weeks. Not more than 75 µg of 99mTc-maraciclatide will be administered intravenously with an activity as close as possible to 740 MBq. Static whole-body imaging will be undertaken after a maximum of 2 hours with further dedicated views of the hands and feet. Total image acquisition time will be approximately 30 minutes. Images will be scored by quantitative and semi-quantitative methods by a blinded observer.

SUMMARY:
The goal of this observational study is to investigate whether 99mTc-maraciclatide imaging prior to biologic therapy tapering and after 3 months can predict those at risk of Rheumatoid arthritis flare.

Participants undergoing routine tapering of biologic drug therapy will have 99mTc-maraciclatide imaging in addition to normal ultrasound imaging and then followed up over 12 months to assess whether an interval scan alone or in combination with the baseline scan is predictive of flare.

DETAILED DESCRIPTION:
Rheumatoid arthritis is a chronic inflammatory condition affecting the joints which over time can cause progressive arthritis and disability. Since the introduction of widespread us of targeted biologic therapies. More patients are now maintained in remission and low disease activity with better long-term outcomes. Making treatment decisions can be challenging as disease activity scores do not always reflect inflammatory disease activity and active inflammation may be present but not manifested by clinically obvious swelling. Ultrasound, and in particular power Doppler (PD), has been shown to be a more sensitive indicator of active inflammatory disease and is widely used in clinical practice to inform decision making.

However, ultrasound is time consuming and thus expensive and it is impractical to image more than a few joints routinely. We have shown that 99mTc-maraciclatide, a nuclear imaging agent that uses equipment routinely available in hospitals, correlates with PD and hence has potential as an accessible, more cost effective and, as is has the potential to image all the joints in a single acquisition, more clinically informative alternative.

Many patients on biologic therapy achieve low disease activity and may be suitable for tapering of medication. This has the advantage of reducing exposure to immunosuppressive medication and reducing costs. Whilst many patients can be tapered safely it is not always clear who is at risk of flaring. It is known that the presence of PD signal can predict higher risk, but this is not routinely used in practice for the reasons above. In this study we will investigate whether 99mTc-maraciclatide imaging prior to tapering and after 3 months can predict those at risk of flare. Success will indicate that it could be used in clinical practice with potential to minimise exposure to unnecessary treatment whilst preserving clinical outcomes, improving patient experience and reducing costs.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of RA according to American College of Rheumatology/EULAR criteria.
2. Clinical remission or LDA and deemed suitable for treatment tapering by their supervising rheumatologist.
3. Existing TNF inhibitor therapy (adalimumab, etanercept, certolizumab pegol, golimumab, infliximab) administered at doses and dosing intervals that have been stable for ≥ 6 months.
4. Aged between 18 and 80 years of age

Exclusion Criteria:

1. Recently received IM/IA steroids (12 weeks washout required).
2. The subject was previously entered into this study or has participated in any other investigational drug or medical device study within 30 days of enrolment.
3. The subject has known allergies to maraciclatide or any constituent of its injectate.
4. The subject size or weight is not compatible with imaging as determined by the investigator.
5. The subject has received any radiopharmaceutical within 7 days or 10 half-lives prior to the imaging day (Day 0).
6. The subject is pregnant or lactating.
7. The subject has severe renal dysfunction, with estimated glomerular filtration rate (eGFR) <30 ml/min/1.73m2.
8. The subject has hepatic insufficiency as demonstrated by ALT (alanine aminotransferase [SGPT]) or AST (aspartate aminotransferase [SGOT]) >3 times the upper limit of normal.
9. The subject presents with any other clinically active, serious, life-threatening disease with a life expectancy of less than 12 months or where participation in the study might compromise the management of the subject or other reason that in the judgment of the investigator(s) makes the subject unsuitable for participation in the study.
10. The subject is claustrophobic or has a movement disorder that prevents him/her from lying still in a supine position for up to 20 minutes at a time.
11. Patients who are currently involved in interventional trials will not be suitable

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: RA patients selected for treatment tapering
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
99mTc-maraciclatide is predictive of risk of flare | 12 months
  Number of patients who flare within 12 months which also have increased 99mTc-maraciclatide

SECONDARY OUTCOMES:
Interval and Baseline scan | 12 months
  Correlations between interval scan scoring alone or in combination with the baseline scan scoring and incidence of flare
Ultrasound correlation | 12 months
  Correlation between ultrasound (grey scale and power Doppler) and 99mTc-maraciclatide scoring at the whole patient and individual joint level
Serological correlation | 12 months
  Correlation between 99mTc-maraciclatide imaging and clinical and serological markers of disease activity

IPD SHARING:
Plan to Share IPD: No